CLINICAL TRIAL: NCT06470919
Title: The Next Generation Vaccine Card: Innovative Technology to Improve Vaccine Equity in Rural and Urban Settings in East Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: African Population and Health Research Center (Other)
Responsible Party: Principal Investigator, Emily Treleaven, Research Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00237101
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Vaccines
Keywords: Kenya; Uganda; Vaccine coverage; Vaccine completion; Vaccine timeliness; Digital health interventions

STUDY DESIGN:
Intervention Model Description: Mothers will be randomized to receive the digital vaccine card access with short message service (SMS) reminders versus mothers who did not receive digital vaccine card access with SMS reminders (treatment/control).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Next Generation digital vaccine card with SMS reminders for upcoming vaccination(s) (Experimental)
  Interventions: Other: SMS reminders for upcoming vaccination(s)
- Pre-intervention cohort (No Intervention): This group will be compared to the post-intervention group to assess the digital vaccine card.

INTERVENTIONS:
Other: SMS reminders for upcoming vaccination(s) — All parents/caregivers of children in participating villages will receive access to a digital vaccine card. This will be used for record-keeping application (digital vaccine registry). Selected parents/caregivers of children will receive SMS messages and reminders related to vaccination.
  Arms: Next Generation digital vaccine card with SMS reminders for upcoming vaccination(s)

SUMMARY:
The research team of investigators from University of Michigan and the African Population and Health Research Center will implement and evaluate a newly-developed digital vaccine card and accompanying mobile application and electronic immunization registry. This will take place in rural Uganda and urban Kenya Health and Demographic Surveillance Systems (HDSS) and the study team will analyze its feasibility, impacts, cost through process, and economic evaluations. The study team will also assess the data quality and equity of the digital vaccine registry and card system.

DETAILED DESCRIPTION:
This study design has three parts or aims for this project, however, only the third aim is considered to be the trial portion and is included in this registration.

ELIGIBILITY:
Inclusion Criteria:

* 1 day to 24 months old

Exclusion Criteria:

* Sites not included in the study

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3522 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Diphtheria, pertussis, and tetanus first dose (DPT1) coverage | 18 months of the intervention period
  Percent (%) of all children born in the intervention period that received the first dose of DPT vaccine (Continuous measure, 0-100%).
Diphtheria, pertussis, and tetanus first dose (DPT3) coverage | 15 months of the intervention period (last 15 months of the intervention period)
  Percent of all children born in the first 15 months of the intervention period that received the third dose of DPT vaccine (Continuous measure, 0-100%).
Dropout rate from DPT1 to DPT3 | 15 months of the intervention period (last 15 months of the intervention period)
  Difference in the proportion of children born in the first 15 months of the intervention period that received the first and third doses of the DPT vaccine (Continuous measure, 0-100%)

SECONDARY OUTCOMES:
Bacillus Calmette-Guerin (BCG) coverage | 18 months of the intervention period (full intervention period)
  Percent of all children born in the intervention period that received the BCG vaccine (Continuous measure, 0-100%).
Measles coverage | 9 months of the intervention period (second half of the intervention)
  Percent of all children born in the first 9 months of the intervention period that received the Measles vaccine (Continuous measure, 0-100%).
Completion of basic immunizations | 9 months of the intervention period (second half of the intervention)
  Percent of all children born in the first 9 months of the intervention period that received all basic recommended immunizations (BCG, oral polio vaccine (OPV), DPT1, DPT2, DPT3, OPV1, OPV2, OPV3, Pneumococcal Conjugate (PCV)1, PCV2, PCV3, rotavirus (Rota)1, Rota2, Rota3, Measles)
Dropout rate from DPT1 to Measles | 9 months of the intervention period (second half of the intervention)
  Difference in the proportion of children born in first 9 months of the intervention period that received the first dose of the DPT vaccine and the Measles vaccine (Continuous measure, 0-100%)
Timeliness of BCG vaccination | 18 months of the intervention period (full intervention period)
  Percent of all children born in the intervention period that received the BCG vaccine by 4 weeks (Continuous measure, 0-100%).
Timeliness of DPT1 vaccination | 15 months of the intervention period (last 15 months of the intervention period)
  Percent of all children born in the intervention period that received the first dose of DPT vaccine by 10 weeks (Continuous measure, 0-100%).
Timeliness of DPT3 vaccination | 15 months of the intervention period (last 15 months of the intervention period)
  Percent of all children born in the intervention period that received the third dose of DPT vaccine by 18 weeks (Continuous measure, 0-100%).
Timeliness of Measles vaccination | 9 months of the intervention period (second half of the intervention)
  Percent of all children born in the intervention period that received the Measles vaccine by 10 months (Continuous measure, 0-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Treleaven, PhD, MPH, Principal Investigator — University of Michigan; Gershim Asiki, MBChB, MSc, PhD, Principal Investigator — African Population and Health Research Center
Locations (2):
- African Population and Health Reseach Center, Nairobi, Kenya, Kenya
- Uganda Christian University, Kasese, Uganda, Uganda

IPD SHARING:
Plan to Share IPD: No